CLINICAL TRIAL: NCT04902534
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose Escalation Safety, Tolerability, and Pharmacokinetic Phase I Clinical Study of Naoqingzhiming Tablets in Chinese Healthy Subjects
Brief Title: Clinical Trial of Naoqingzhiming Tablets in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GX-SGJG-001
Record Dates: First submitted 2020-09-23; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, single dose and multiple dose escalation phase I clinical study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naoqingzhiming Tablets (Experimental): Naoqingzhiming Tablets, specification:500mg(contains echinacoside 180mg) Single dose ascending. Qualified subjects will enter 6 dose groups in order from low to high: 180mg, 360mg, 720mg, 1080mg, 1620mg and 2160mg, with increasing dose design The first group (180mg) is a pre-experiment. Two subjects were selected and all received the test drug.
  Groups 2 to 6 received the experimental drug in 8 patients per group. Multi-dose ascending was divided into two groups: 360mg and 720mg. 10 subjects in each group received the test drug 3 times a day for 14 consecutive days.
  Interventions: Drug: Naoqingzhiming Tablets (contains echinacoside 180mg)
- placebo (without active ingredients echinoside) (Placebo Comparator): Placebo Tablets, specification: 500mg(without echinoside) Single dose. Groups 2 to 6 received the placebo in 2 patients per group. Multi-dose ascending. Two people in each group received placebo 3 times a day for 14 consecutive days.
  Interventions: Drug: placebo of Naoqingzhiming Tablets (without echinacoside)

INTERVENTIONS:
Drug: Naoqingzhiming Tablets (contains echinacoside 180mg) — Single dose escalation and multiple dose escalation
  Arms: Naoqingzhiming Tablets
Drug: placebo of Naoqingzhiming Tablets (without echinacoside) — Single dose escalation and multiple dose escalation
  Arms: placebo (without active ingredients echinoside)

SUMMARY:
A single-center, randomized, double-blind, placebo-controlled, dose escalation safety, tolerability, and pharmacokinetic phase I clinical study of Naoqingzhiming Tablets in Chinese healthy subjects.

DETAILED DESCRIPTION:
The single-dose trial plan enrolls 52 Chinese healthy subjects. Qualified subjects will enter 6 dose groups in order from low to high: 180mg, 360mg, 720mg, 1080mg, 1620mg and 2160mg, with increasing dose design The first group (180mg) is a pre-test. Two subjects were selected and all received the test drug. They were observed for 24 hours after a single dose for safety assessment, and followed up 7-10 days after leaving the group or early withdrawal. If more than one subject has an adverse event that meets CTCAE V5.0 Grade II or above and is judged to be related to the test drug, then consider reducing the dose, otherwise proceed to the next dose group trial. Groups 2, 3, 4, 5, and 6 follow the "8+2 principle", with 10 subjects in each group, 8 receive the test drug, and 2 receive the placebo. Observe for 24 hours after a single dose for safety assessment , And follow up 7-10 days after leaving the group or early withdrawal. Each subject received only one dose group of the trial, only one study drug (experimental drug or placebo), and no longer participated in the other dose group trials or took two study drugs. During the dose escalation process, after completing the safety assessment of the previous dose group, if the dose escalation suspension standard is not met, continue the test of the lower-dose group. It is not allowed to conduct the test of 2 or more dose groups at the same time. In the above six groups of trials, it is not only necessary to observe the safety and tolerability of the subjects taking the study drug, but also to evaluate the pharmacokinetic characteristics of a single dose.

According to the results of animal pharmacokinetic studies, the dose grouping for the multiple-dose study is tentatively set to 2 groups: 360mg group and 720mg group.

The multiple-dose study plan recruited 24 Chinese healthy subjects, following the "10+2 principle", each group of 12 subjects, 10 cases received the test drug, 2 cases received placebo, 3 times a day, continuous medication On 14 days, continue to observe for 24 hours after the last administration for safety assessment, and follow up 7-10 days after leaving the group or early withdrawal. In the process of continuous medication, if 3/10 and more than 3/10 of the subjects in a dose group who received the test drug withdraw from the trial due to adverse events related to the test drug, the trial should be aborted; after completing the first group, it is safe After the sexual assessment, if the suspension criteria are not met, the second group of trials will continue. Each subject only participates in one group of trials and only receives one study drug (experimental drug or placebo), and no longer participates in other group trials or takes two study drugs. In the above two groups of trials, it is not only necessary to observe the safety and tolerability of multiple administrations, but also to evaluate the pharmacokinetic characteristics of multiple administrations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects understand well trial purpose, nature, content, process and possible adverse reactions, and voluntarily sign an informed consent form.
* Healthy male or female aged between 18 and 65 years old (including the critical value).
* The body mass index is in the range of 19-26kg/m2 (including the critical value). The weight of male is not less than 50 kg, and that of female is not less than 45 kg (including the critical value).
* Subjects who had not any medical history of cardiovascular, digestive, respiratory, nervous, haemal diseases or hepatic/renal impairment.The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: physical examination, 12-lead ECG, vital sign measurements, Chest X-ray, abdominal ultrasound and laboratory safety tests .
* The subjects have no family planning within 6 months and could select contraceptive method. They have no sperm and egg donation program.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.
* The subjects could communicate well with researchers and complete the study according to the protocol.

Exclusion Criteria:

* Any history of hypersensitivity or idiosyncratic reactions to any food or drug, especially for drugs containing echinacoside.
* Hepatitis (including hepatitis B and C), positive screening results for AIDS or syphilis;
* ALT or/and AST or/and TBIL ≤1.5 times the upper limit of normal Cr,BUN≥upper limit of normal, or Ccr≤80mL/min.
* Any history of acute or chronic illness that might affect drug absorption, and/or metabolism;
* Any history of drug abuse in the past 6 months or drug use 3 months prior to screening;
* Any history of alcohol abuse 3 months prior to screening or moderate drinkers (drink more 2 units per day or 14 units per week);
* Smoking more than 5 cigarettes per day during the 3 months prior to screening;
* Blood donation, massive blood loss (#400mL) or enrolled in other clinical trials 3 months prior to screening;
* Any use of other prescription drugs (including contraceptive)、over-the-counter drugs, Chinese herbal medicine, health care products and 14 days prior to medication for this study;
* Any use of prescription or over-the-counter drugs, functional vitamin, herbal/ alcohol products, grapefruit-containing or caffeine/xanthine-rich food and beverages 48 h prior to medication for this study;
* Dysphagia or having special dietary requirements;
* Occurring acute disease in the screening period or before the medication;
* Lactating or pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 500 days
  Maximum tolerated dose for a single dose
Occurrence rate of Adverse Events | 500 days
  Adverse events were recorded to evaluate the safety of the studied drugs

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 500 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 500 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 500 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Beijing Sili'an Pharmaceutical Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor.